CLINICAL TRIAL: NCT03429881
Title: Microparticle Generation After Laparoscopic Surgical Treatment for Endometrioma: a Pilot, Prospective, Randomized Study Comparing Stripping With CO2 Laser Vaporization
Brief Title: Microparticle Generation After Laparoscopic Surgical Treatment for Endometrioma.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Francisco Carmona (Other)
Responsible Party: Sponsor-Investigator, Francisco Carmona, Professor, Hospital Clinic of Barcelona
Organization: Hospital Clinic of Barcelona (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: HCB/2015/0068
Record Dates: First submitted 2018-02-05; First posted 2018-02-12 (Actual); Last update posted 2018-02-12 (Actual); Status verified 2018-02

CONDITIONS: Microparticle; Endometriosis; Laparoscopy
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laparoscopic stripping ovarian endometriomas (Active Comparator)
  Interventions: Procedure: Stripping versus laser CO2
- Laser CO2 treatment ovarian endometriomas (Active Comparator)
  Interventions: Procedure: Stripping versus laser CO2

INTERVENTIONS:
Procedure: Stripping versus laser CO2 — Patients were randomly selected to undergo either CO2 laser vaporization (L group) or laparoscopic stripping (S group) of OE.

SUMMARY:
Study objective: To evaluate serial generation of microparticles (MPs) after laparoscopic stripping or CO2 laser vaporization in surgical treatment of patients with ovarian endometrioma (OE).

Design: A prospective, randomized, blinded, pilot study, including 33 patients. Setting: Tertiary university hospital from April 2015 to June 2017. Patients: 33 women with unilateral OE undergoing laparoscopic surgery. Intervention: Patients were randomly selected to undergo either CO2 laser vaporization (L group) or laparoscopic stripping (S group) of OE.

Measurements and Main results: Blood samples were collected before surgery, and at 2 hours, 24 hours, 1 month, and 3 months after surgery. MPs generation curve after ovarian endometrioma surgery was performed.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 40 years and unilateral symptomatic OEs ≥3 cm.

Exclusion Criteria:

* previous pelvic surgery, history of cancer, suspected malignancy, presurgical suspicion or evidence of deep endometriosis, presurgical suspicion or evidence of premature ovarian failure, and the use of estrogen suppressive drugs, including oral contraceptives, GnRH-agonists, progestins, or danazol in the preceding 3 months. We excluded patients with suspicion of deep endometriosis according to an extensive preoperative work-up (including magnetic resonance imaging when necessary) routinely performed in such patients.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2018-02-05 (Actual); Primary Completion 2018-02-05 (Actual); Study Completion 2018-02-05 (Actual)

PRIMARY OUTCOMES:
Microparticle levels after two laparoscopic treatments of ovarian endometriomas | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clinic, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
Publication in an indexed journal
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Within 2018